CLINICAL TRIAL: NCT00844142
Title: Randomized Controlled 12 Months Trial With Etanercept (Enbrel ®) vs. Sulfasalazine in Early Axial Spondyloarthritis With Focus on Improvement of Acute Inflammatory Lesions as Detected by MRI. Amendment 4: 1-Year Extension of Study
Brief Title: Enbrel-Sulfasalazin-Early-Axial Spondyloarthritis (AS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Prof. Dr. med. Joachim Sieper, Charité Rheumatology Campus Benjamin-Franklin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M01; Enbrel-Sulfa-Early-AS
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Moderate to Severe Active Axial Spondyloarthritis
Keywords: ankylosing spondylitis; axial spondyloarthritis; magnetic resonance imaging; etanercept; sulfasalazine
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis | interventions — Etanercept; Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): etanercept 25mg twice weekly
  Interventions: Drug: Etanercept 25mg
- 2 (Active Comparator): Sulfasalazine 2000- 3000mg daily
  Interventions: Drug: Sulfasalazine

INTERVENTIONS:
Drug: Etanercept 25mg — patients will receive etanercept 25mg twice weekly
  Arms: 1
Drug: Sulfasalazine — in this arm patients will receive sulfasalazine 2000- 3000mg per os daily
  Arms: 2

SUMMARY:
Efficacy - To assess efficacy of etanercept versus sulfasalazine when added to NSAIDs in patients with moderate to severe active early axial spondyloarthritis duration of ongoing axial symptoms of less than 5 years. Primary outcome is change of active inflammatory lesions in sacroiliac joints and spine as detected by MRI at 12 months. Secondary outcome parameters are clinical and laboratory efficacy parameters and MRI changes at 6 months and 2 years. Comparisons will be made within the two treatment arms and compared to baseline. At the 1 year extension phase comparisons will be also made between year 1 and year 2. At the end of the extended study a pelvic x-ray is planned.

DETAILED DESCRIPTION:
Randomized controlled study with two treatment arms (Phase II), 1 year open extension

Efficacy - To assess efficacy of etanercept vs. sulfasalazine when added to NSAIDs in patients with moderate to severe active early axial spondyloarthritis duration of ongoing axial symptoms of less than 5 years. Primary outcome is change of active inflammatory lesions in sacroiliac joints and spine as detected by MRI at 12 months. Secondary outcome parameters are clinical and laboratory efficacy parameters and MRI changes at 6 months and 2 years. Comparisons will be made within the two treatment arms and compared to baseline. At the 1 year extension phase comparisons will be also made between year 1 and year 2. At the end of the extended study a pelvic x-ray is planned. For etanercept group: To assess whether etanercept will show sustained long term response over 1 more year. To assess whether etanercept will slow or stop progression as shown by MRI.For sulfasalazine group: to assess whether etanercept will show long term response over 1 year. To assess whether etanercept will slow or stop progression as shown by MRI. For all patients who are in remission the duration of remission will be assessed for a maximum of one year. In case of a flare of the disease these patients will be (re-) treated with etanercept and efficacy will be assessed. Safety - To study the long-term safety of etanercept in patients with moderate to severe active early axial spondyloarthritis compared to patients treated with sulfasalazine over a period of one year.

Patients will be treated for 1 year either with etanercept 2x25mg per week subcutaneously or with sulfasalazine 2g/ day given orally. Following screening and baseline evaluations, patients will be assessed at week 2, 4, 6, 8, 10, 12, 24, 36 and 48. Efficacy and safety measurements will be recorded throughout the entire study. The study will be followed by a 60 weeks follow-up phase after week 48 (end of treatment phase). In case of flare they will be (re-)treated with etanercept for further 60 weeks (until week 108). All patients from the former etanercept group who are not in remission will continue to be treated with etanercept for 60 weeks (weeks 60, 72, 84, 96, 108). All patients from the former sulfasalazine group who are not in remission will be switched to etanercept for 60 weeks (at weeks 50, 54, 60, 72, 84, 96, 108).

Treatment arms:Arm 1: 40 patients receive etanercept 2x25 mg weekly subcutaneous injectionArm 2: 40 patients receive sulfasalazine up to 2 g/day (up to 3 g/ per day)

Duration of the study:12 months. For patients in remission a 12 months follow up period will be enclosed. Treatment will be continued for patients in case of flare or in patients who did not achieve remission for 60 weeks. The study is planned start at September 2005. Patients will be recruited over a 12 months period. Altogether the duration of the study is up to 51 months. All patients who are willing to participate in the extension will be treated for another 60 weeks.

Patient Population:Only active axial SpA patients with a disease duration (measured from time of ongoing spinal symptoms) of less than 5 years will be included. This implies that patients with both radiological evidence of sacroiliitis (fulfilling the modified New York criteria for AS) and without radiological evidence of sacroiliitis (see inclusion criteria) will be included.

Efficacy Variables:Primary endpoint:· Reduction of active inflammatory lesions in MRI at 12 monthsSecondary endpoints:

* ASAS 20%, 40%, 70% response, ASAS criteria for partial remission· BASDAI 20%, 50%, 70% improvement · BASFI · Mobility examinations: BASMI, Chest Wall Expansion· disease controlling antirheumatic therapy criteria (DC-ART20) (5 out of 6)*· CRP, ESR· Quality of Life: SF-36· Numeric Rating Scale (NRS) - physicians global, patients global, general pain, nocturnal pain · Enthesitis index (Maastricht scale)· swollen joint count· EQ-5D· Socio-economic questionnaire· Chronic changes in MRI at 6, 12 months and 108 weeks· Reduction of active inflammatory lesions in MRI at 6 months and chronic lesions at 6 and 12 months and 108 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 50 years of age who have moderate to severe active axial spondyloarthritis.
* Diagnosis made by :Chronic low back pain (duration > 3 months, onset < 45 years of age)plus 3 out of the 6 following criteria if imaging is positive or 4 out of the following 6 criteria if imaging is negative ·
* Inflammatory back pain:

  * Good or very good response to NSAIDs
  * One or more of the following extraspinal manifestations: uveitis, peripheral arthritis, enthesitis, HLA-B27 positive
  * Positive imaging: MRI showing acute inflammatory lesions in spine or SIJ (in the past) or bilateral sacroiliitis grade 2-4 or unilateral sacroiliitis grade 3-4 in x-ray not older than 12 months
  * Positive family history for SpA
  * MRI at screening showing acute inflammatory lesions in SIJ or spine
* Active disease is defined as:

  * a BASDAI score of >=4
  * back pain score (BASDAI question 2) of >= 4 despite concurrent NSAID therapy, or intolerance to NSAIDs.
* Other inclusion criteria include, if on prednisone:

  * <7.5 mg per day
  * stable for 4 weeks prior to baseline
* Women of child bearing potential must have a negative pregnancy test at study baseline and use an adequate, effective method of contraception for a duration of 6 months after stop of etanercept therapy. Sexual active men must use an accepted method of contraception for a duration of 6 months after stop of etanercept therapy.
* Reading a normal chest/lung x-ray which should have been performed within the last 12 weeks before inclusion
* Able to self-administer injectable drug supplies or have a caregiver who will do so.
* Able to store injectable test article at 2° to 8° C.

Exclusion Criteria:

* Disease duration of longer than 5 years
* History of active tuberculosis (TB), histoplasmosis or listeriosis.
* History of positive HIV status, known hepatitis B or C
* History of malignancy other than carcinoma in situ of the cervix or adequately treated non-metastatic squamous or basal cell skin carcinoma.
* Antibiotic treatment within 3 weeks prior to screening.
* Previous treatment with TNF-alpha blockers
* Treatment with sulasalazine in the last 6 months before participation in the clinical trial
* severe internal medical diseases such as severe cardiac, hepatic, gastrointestinal, neurological, psychiatric diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-11; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Reduction of active inflammatory lesions in MRI at 12 months. | 108 weeks

SECONDARY OUTCOMES:
Secondary outcome: ASAS 20%, 40%, 70% response, ASAS criteria for partial remission· BASDAI 20%, 50%, 70% improvement · BASFI · | 108 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, MD, Principal Investigator — Charite, Campus Benjamin-Franklin, Rheumatology, Berlin, Germany
Locations (9):
- Germany (9):
  - Charité Campus Mitte, Rheumatology, Berlin
  - Praxis Mielke, Berlin
  - Praxis Zinke, Berlin
  - Klinikum Buch, Berlin
  - Waldkrankenhaus, Berlin
  - Schlossparkklinik, Rheumatology, Berlin
  - Immanuel Krankenhaus, Berlin
  - Praxis Klopsch, Neubrandenburg
  - Praxis Bohl-Bühler, Potsdam

REFERENCES:
- [Derived] Torgutalp M, Rademacher J, Proft F, Hermann KG, Althoff C, Haibel H, Protopopov M, Sieper J, Rios Rodriguez V, Poddubnyy D. Association between resolution of MRI-detected inflammation and improved clinical outcomes in axial spondyloarthritis under long-term anti-TNF therapy. RMD Open. 2025 Jan 6;11(1):e004921. doi: 10.1136/rmdopen-2024-004921. PMID 39762123
- [Derived] Song IH, Hermann KG, Haibel H, Althoff CE, Poddubnyy D, Listing J, Weiss A, Lange E, Freundlich B, Rudwaleit M, Sieper J. Prevention of new osteitis on magnetic resonance imaging in patients with early axial spondyloarthritis during 3 years of continuous treatment with etanercept: data of the ESTHER trial. Rheumatology (Oxford). 2015 Feb;54(2):257-61. doi: 10.1093/rheumatology/keu263. Epub 2014 Aug 19. PMID 25140041
- [Derived] Song IH, Hermann KG, Haibel H, Althoff CE, Poddubnyy D, Listing J, Weiss A, Buss B, Freundlich B, Lange E, Alten R, Rudwaleit M, Sieper J. Consistently Good clinical response in patients with early axial spondyloarthritis after 3 years of continuous treatment with etanercept: longterm data of the ESTHER trial. J Rheumatol. 2014 Oct;41(10):2034-40. doi: 10.3899/jrheum.140056. Epub 2014 Jul 15. PMID 25028375
- [Derived] Weiss A, Song IH, Haibel H, Listing J, Sieper J. Good correlation between changes in objective and subjective signs of inflammation in patients with short- but not long duration of axial spondyloarthritis treated with tumor necrosis factor-blockers. Arthritis Res Ther. 2014 Jan 30;16(1):R35. doi: 10.1186/ar4464. PMID 24476416